CLINICAL TRIAL: NCT03771365
Title: An International Multi-center Prospective Cohort Study Comparing the Safety and Efficacy of Super-mini-PCNL, Mini-PCNL and Standard PCNL in the Treatment of ≥2cm Renal Stones
Brief Title: Standard-PCNL vs Mini-PCNL vs Super-mini PCNL for the Treatment of ≥2 cm Renal Stone
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Military Medical Academy, Bulgaria (Other); Massachusetts General Hospital (Other); Hospital de Clinicas José de San Martín (Other); Goldstadt Private Clinic (Unknown); University College London Hospitals (Other); Hospital de Base do Distrito Federal (Unknown); Mexican National Council of Urology (Unknown); Vancouver General Hospital (Other); Lions Kidney Hospital and Urology Institute (Unknown); Mt. Carmel Diocesan General Hospital (Unknown); Clinical Emergency County Hospital (Unknown); University of Belgrade (Other); Hospital das Clínicas, University of Sao Paulo Medical School (Unknown); Vayodha and Venus International Hospitals (Unknown); University Hospital of Vinalopo (Unknown); Sismanoglio General Hospital (Other); New Mowasat Hospital (Unknown)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 1stAHGZMU
Record Dates: First submitted 2018-11-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Stone, Kidney; Lithiasis Renal; Surgery
Keywords: percutaneous nephrostolithotomy; renal stone; safety; efficacy
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard-PCNL: Perform PCNL with ≥24 Fr access tract for the treatment of ≥2 renal stones
  Interventions: Procedure: Standard-PCNL
- Mini-PCNL: Perform PCNL with 12-20 Fr access tract for the treatment of ≥2 renal stones
  Interventions: Procedure: Mini-PCNL
- Super-mini PCNL: Perform SMP for the treatment of ≥2 renal stones
  Interventions: Procedure: SMP

INTERVENTIONS:
Procedure: Standard-PCNL — percutaneous nephrostolithotomy (PCNL) with ≥24 Fr access tract for the treatment of ≥2 cm renal stone
  Groups: Standard-PCNL
Procedure: Mini-PCNL — percutaneous nephrostolithotomy (PCNL) with 12-20 Fr access tract for the treatment of ≥2 cm renal stone
  Groups: Mini-PCNL
Procedure: SMP — percutaneous nephrostolithotomy (PCNL) with 10-14 Fr access tract for the treatment of ≥2 cm renal stone
  Groups: Super-mini PCNL

SUMMARY:
Background: Standard-PCNL was considered as the first choice for ≥2 cm renal stones. Miniaturized technique Mini-PCNL has also been implicated in the past two decades. Recently, Super-mini PCNL (SMP) was introduced to treated ≤2.5cm renal stone. The miniaturized techniques seemed to take a longer operating time and have risk of getting infectious complications. However, there is no high quality of evidence showing that which kind of PCNL is best or what kind of patients is suitable for standard-PCNL, mini-PCNL or SMP.

Objective: To compare the efficacy and safety of Standard-PCNL (≥24Fr), Mini-PCNL (12-20Fr) and SMP(10-14Fr) for the treatment of ≥2 cm renal stones Study design: This study is a prospective, observational, international, multicenter registry cohort study Study population: All patients ≥14 years with ≥2 cm renal stone who are planned for Standard-PCNL, Mini-PCNL or SMP are eligible for this study.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Percutaneous nephrolithotomy (PCNL) is the first-choice for the treatment of renal stone ≥20 mm with high stone free rate (SFR). However, there are some sever complications such as bleeding. Severe bleeding needs arterial embolization, which might impair the renal function. The size of percutaneous access tract has been proven to be closely related to the risk of bleeding complications. Mini-PCNL was firstly introduced by Jackman in 1998 to treat pediatric renal stone with the aim to lower the morbidity. Mini-PCNL was gradually applied to adults. In recent years, urologists were still attempting to reduce size of the sheath and modify the sheath. They aimed to reduce the risk of bleeding. The first generation SMP consists of a 10-14 F access sheath with a suction-evacuation function and a 7-F nephroscope with enhanced irrigation was introduced by Guohua Zeng's group in 2014. In 2016, Guohua Zeng's group continued to introduce a modified SMP technique and system. The most remarkable feature of the new generation super-mini percutaneous nephrolithotomy (New-SMP) was metal irrigation-suction sheath which made the new system have higher efficiency than the old one. With the modified SMP technique and system, SMP was performed to treat large renal stone. (≥2cm). Moreover, SMP with an irrigation-suction sheath obviously improved the efficiency of removing the fragments and lower the intrapelvic pressure.

Although miniaturized techniques decreased the bleeding-related morbidity and have a similar SFR, they seemed to take a longer operating time and have risk of getting infectious complications. However, till now, no high quality of evidence demonstrated that what size of tract is the best for the treatment of ≥2 cm renal stone. Perhaps the investigators should find out a subgroup suitable for standard-PCNL, Mini-PCNL or SMP respectively.

STUDY OBJECTIVES The aim of this registry is to review current clinical practice on PCNL for stone treatment. The investigators will explore the answers to the following questions: What kind of PCNL urologists prefers to used? Is there a best cutoff based on the size of stones to divide the patients into subgroups, or a scoring system to decide which kind of PCNL is the best choice for individuals? Primary Objective To compare the stone free rate (SFR) (%) among standard-PCNL, Mini-PCNL and SMP for the treatment of ≥2 cm renal stone.

Secondary Objectives

1. Bleeding complication: hematocrit drop (g/L) and rate of transfusion (%).
2. Infectious complication: rate of getting fever (≥38℃) (%) and urosepsis (%).
3. Intraoperative indexes: operating time (mins), rate of tubeless/total tubeless (%).
4. Postoperative indexes: hospital stay (mins), visual analogue scale (VAS) score (range from 0-10, the higher value represents the worse outcome) STUDY DESIGN This study is a prospective, observational, international, multicenter registry cohort study SELECTION AND ENROLLMENT OF PARTICIPANTS Clinical Recruitment All sites for this pilot study are recruited by IAU Members. Each participating center should obtain ethical approval, as needed, according to local regulations.

Each participating centre will include all consecutive eligible patients. PCNL procedures are performed according local protocols and surgeons' own propensity. Data will be collected in the IAU online platform (http://47.74.212.47/#/login), which is developed by IAU. Each participating center has own account and password to login and collect data. Data analysis will be coordinated by IAU.

Study Population All patients ≥14 years with ≥2 cm renal stone who are planned for Standard-PCNL, Mini-PCNL or SMP are eligible for this study.

Surgical procedure The procedure of SMP, mini-PCNL and Standard-PCNL was according to surgeons' propensity, the related details were recorded online.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥14 years old
* Patient is a candidate for Standard-PCNL, Mini-PCNL or SMP treatment of a renal stone

Exclusion Criteria:

* Patient <14 years old

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients ≥14 years with ≥2 cm renal stone who are planned for Standard-PCNL, Mini-PCNL or SMP are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate (SFR) (%) | 1-3 months after the day of DJ stent/ureteral catheter removal or the day of operation (if no DJ stent or ureteral catheter placed postoperatively).
  Stone free rate (SFR) (%) are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 4mm, asymptomatic, non-obstructive and non-infectious stone particles.

SECONDARY OUTCOMES:
Perioperative complications | intraoperatively or ≤ 1 month postoperatively
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: Undecided
It is a international multi-center prospective cohort study, the data is not available to other researchers before the agreement from all the centers